CLINICAL TRIAL: NCT04075916
Title: A Trial of Transplanting Hepatitis C Kidneys Into Hepatitis C-Negative Kidney Recipients
Acronym: THINKER-NEXT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Gilead Sciences (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10067385; U01DK126654 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epclusa (sofosbuvir/velpatasvir) (Experimental): Epclusa is taken by mouth for 12 weeks as per the FDA label.
  Interventions: Drug: Epclusa

INTERVENTIONS:
Drug: Epclusa — All patients will receive 12 weeks of sofosbuvir/velpatasvir as per the FDA label.

SUMMARY:
The Transplanting Hepatitis C Kidneys into Negative KidnEy Recipients [THINKER-NEXT] study will include adult kidney transplant candidates without hepatitis C virus (HCV) infection on the transplant waiting list who will consent to kidney transplantation from a deceased donor infected with HCV, followed by treatment with a direct acting antiviral. The one-year allograft function and one-year risk of CMV infection will be compared between THINKER-NEXT kidney transplant recipients and matched recipients who received hepatitis C uninfected kidney transplants (these patients are called Transplant Cohort). The survival rate of patients opting-in for offers of kidneys from HCV-viremic donors will be compared to the survival rate of matched comparators from the kidney transplant waitlist who did not consent to receive offers of a HCV-viremic kidney. Lastly, renal pathologic findings will be compared among HCV-viremic donors and HCV-negative comparator donors.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Active waiting list status for isolated kidney transplant
* 18 years of age or older
* No living kidney donor
* Panel reactive antibody (PRA) ≤97% (most recent cPRA at time of screening). Patients with a PRA of 98-100% at screening can be included unless patient has a most recent cytotoxic PRA of >25% or calculated PRA >50% where multiple moderate level HLA antibodies exist and in the opinion of the local site investigator represents substantial HLA sensitization. If patient has a PRA of 98-100%, the donor-recipient pair must meet additional eligibility criteria.

Exclusion Criteria:

* Hepatocellular carcinoma
* Hepatitis B surface antigen and/or DNA positive
* Active Hepatitis C infection
* HIV RNA-positive or HIV antibody positive
* Other chronic liver disease (excluding non-alcoholic fatty liver disease [NAFLD] with normal liver enzymes)
* Persistently elevated liver transaminases (defined as the upper limit of normal at the reference laboratory)
* Advanced hepatic fibrosis or cirrhosis
* Primary Focal Segmental Glomerulosclerosis (FSGS), FSGS recurring in initial transplant, or other disease process at high risk of early graft failure per the treating transplant nephrologist
* Current use of amiodarone or dronedarone (due to interaction with sofosbuvir)
* Transplant candidate requires antibody desensitization protocol for transplantation
* Female who is pregnant, planning to become pregnant during the study, or breast-feeding
* Participation in another interventional study, from a period starting 6 months prior to screening to last study visit, that the study PIs judge would interfere with either the aims or the safety of the THINKER-NEXT study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Post-treatment sustained virologic response (SVR) to direct-acting antiviral (DAA) | Baseline to 24 weeks
  The primary analysis will be based on a calculation of SVR rates (number of subjects with SVR-12; negative HCV RNA 12 weeks after completing Epclusa therapy)/(number of subjects treated with Epclusa post-kidney transplantation)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reese, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - Jackson Memorial Hospital/University of Miami, Miami, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York Presbyterian Hospital/Columbia University, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT04075916/ICF_000.pdf